CLINICAL TRIAL: NCT07343869
Title: Prospective Multicenter Cohort on Esophageal Submucosal Dissection: Evaluation of Technical, Oncological, and Organizational Outcomes in Real-Life Practice
Brief Title: Multicenter Prospective Cohort on Esophageal Endoscopic Submucosal Dissection
Acronym: FEO
Status: Not yet recruiting | Type: Observational
Sponsor: Société Française d'Endoscopie Digestive (Other)
Responsible Party: Principal Investigator, Bertrand Brieau, Principal Investigator, Medical doctor, Société Française d'Endoscopie Digestive
Other Study IDs: SFED-162
Record Dates: First submitted 2025-12-03; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Superficial Esophageal Cancer; Oesophageal Adenocarcinoma; Oesophageal Squamous Cell Carcinoma; Barretts Esophagus With Dysplasia
Keywords: Endoscopic esophageal disection; Endoscopic resection; Endoscopic submucosal dissection; Curative resection
MeSH Terms: conditions — Adenocarcinoma Of Esophagus; Esophageal Squamous Cell Carcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In France in 2018, there were an estimated 2,074 new cases of esophageal adenocarcinoma and 3,224 cases of squamous cell carcinoma. The estimated deaths from esophageal cancer were 3,725, with a standardized 5-year net survival rate of 20% for cases diagnosed between 2010 and 2015, mainly due to late diagnosis.

Surgery was historically the standard treatment for localized disease but carries significant morbidity. Over the past decade, endoscopic treatments, particularly endoscopic submucosal dissection (ESD), have become the reference approach for superficial esophageal cancers.

After endoscopic resection, histological analysis allows classification of recurrence risk into very low, low, and high categories. Predicting lymph node or distant recurrence is complex, depending on factors such as depth of wall infiltration, lymphovascular invasion, and tumor differentiation. The frequent combination of unfavorable histological features may have led to an overestimation of lymph node involvement risk in T1b cancers.

ESD is widely performed in France, with over 1,600 procedures reported in 2023 for esophageal and gastric lesions, demonstrating the feasibility of a large observational study.

This multicenter French cohort will evaluate technical, oncological, and organizational outcomes of esophageal ESD, including overall survival, recurrence-free survival, and management of residual Barrett's esophagus. It will also identify predictive factors for treatment success, recurrence, and complications, providing real-world evidence to guide patient management.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥ 18 years old)
* Patients referred for endoscopic resection of an esophageal lesion and treated by submucosal dissection
* Patients managed in one of the participating centers
* Patient who has received oral and written information about the study and has not objected to participation
* Patients covered by a social security or health insurance scheme.

Exclusion Criteria:

* Patient refusal after reading the information sheet
* Patient under legal protection (guardianship, curatorship, court-ordered protection)
* Inability to inform the patient due to cognitive impairment, language barrier, or medical emergency
* Patients previously included for another lesion in the same study
* Pregnant or breastfeeding women.
* Patient deprived of liberty.
* Patient currently enrolled in another clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible patients include all individuals referred to a participating center for endoscopic resection of an esophageal lesion and treated by submucosal dissection. This is a prospective, multicenter, observational study, conducted on an intention-to-treat basis. All consecutive patients referred for esophageal ESD will be included.
Sampling Method: Non-Probability Sample
Enrollment: 750 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2031-12-01 (Estimated); Study Completion 2036-02-01 (Estimated)

PRIMARY OUTCOMES:
Recurrence-free survival according to adjuvant treatment | From enrollment to 5 years
  Recurrence-free survival will be evaluated in patients after endoscopic submucosal dissection (ESD) of superficial esophageal carcinoma. Patients may receive adjuvant therapy (surgery, chemotherapy, or chemoradiotherapy) at the treating physician's discretion. Recurrence includes local, regional, or metastatic relapse as defined by clinical, endoscopic, and imaging criteria and validated by multidisciplinary team discussion. Recurrence will be monitored throughout the 5-year follow-up period to compare outcomes between patients receiving adjuvant therapy versus surveillance.

SECONDARY OUTCOMES:
R0 resection rate | From ESD to 5 years
  Proportion of patients with tumor-free lateral and deep margins confirmed by histopathology.
En bloc resection rate | From ESD to 5 years
  Proportion of lesions resected in a single piece exclusively by ESD.
Curative resection rate | From ESD to 5 years
  Proportion of R0 resections meeting favorable histological criteria: no lymphovascular invasion, no tumor budding, well-differentiated tumor, submucosal invasion <200 µm (squamous cell carcinoma) or <500 µm (adenocarcinoma).
30-day complication rate | 30 days post-ESD
  Rate of per- or post-procedural bleeding, immediate or delayed perforation, and strictures requiring endoscopic dilation.
Rate of MDTB presentation | From ESD to 5 years
  Proportion of patients whose management was discussed in a multidisciplinary team meeting.
Concordance between MDTB decision and actual management | From ESD to 5 years
  Proportion of patients for whom the implemented management matched the MDTB recommendation.
Rate of patients receiving adjuvant treatment | From enrollment to 5 years
  Proportion of patients receiving any adjuvant therapy after ESD (surgery, radiotherapy, chemotherapy, immunotherapy, etc.).
Rate of complementary Barrett's eradication treatment (radiofrequency or other) | From ESD to 5 years
  Proportion of patients treated for residual Barrett's esophagus using radiofrequency ablation or other endoscopic techniques.
Morbidity of complementary treatments | From ESD to 5 years
  Rate of complications related to adjuvant therapy or Barrett's treatment
Efficacy of complementary treatments | From complementary treatment to 5 years
  Rate of complete remission of intestinal metaplasia or oncologic control following complementary tratmets
Prognostic factors for recurrence (local, regional, metastatic) | From enrollment to 5 years
  Identification of clinical, endoscopic, and histological variables associated with increased risk of recurrence, analyzed using univariate and multivariate methods.
Predictive factors for post-ESD complications | From ESD to 5 years
  Analysis of factors associated with immediate or delayed complications (bleeding, perforation, stenosis) according to patient characteristics, ESD procedure, and adjuvant therapy.
Predictive factors for R0 resection | From ESD to 5 years
  Analysis of clinical, endoscopic, and procedural variables predictive of complete R0 resection.
Diagnostic accuracy of optical endoscopic classifications vs. histology | From ESD to pathology report
  Accuracy of endoscopic optical classifications in predicting histology prior to resection, compared to histopathology results.
Impact of center volume on outcomes | From enrollment to 5 years
  Evaluation of the influence of annual ESD procedure volume in a center on technical and oncologic outcomes

CONTACTS AND LOCATIONS:
Locations (1):
- Jules Verne Clinic, Nantes, France

IPD SHARING:
Plan to Share IPD: Undecided